CLINICAL TRIAL: NCT03777501
Title: The Effect of Whole Body Vibration on Sensorimotor Function in Individuals With Parkinson's Disease
Brief Title: The Effect of Whole Body Vibration in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Kuan-yi Li, Associate professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201702010B0C603
Record Dates: First submitted 2018-12-07; First posted 2018-12-17 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
Keywords: proprioception; vibration; balance
MeSH Terms: conditions — Parkinson Disease | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: randomized double-blinded controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-random whole body vibration group (Experimental): Each participant will receive the non-random type whole body vibration treatment about one hour after the administration of medicine.
  Interventions: Behavioral: non-random whole body vibration
- conventional therapy group (Active Comparator): For the conventional therapy group, participants will receive the occupational therapy including dynamic balance training and functional ambulatory training. Each session is 10 minutes.
  Interventions: Behavioral: occupational therapy

INTERVENTIONS:
Behavioral: non-random whole body vibration — Each participant will receive the treatment about one hour after the administration of medicine. For non-random whole body vibration group, participants will be required to maintain the erect standing position on the vibratory platform and the frequency and amplitude of vibratory stimuli will be 6Hz and 3mm respectively. Each treatment includes five sessions and each session is composed of one minute whole body vibration and one minute rest.
  Arms: non-random whole body vibration group
Behavioral: occupational therapy — Participants will receive the occupational therapy including dynamic balance training and functional ambulatory training.
  Arms: conventional therapy group

SUMMARY:
Previous studies reported that whole body vibration has the potential impact on balance and walking abilities in individuals with Parkinson's disease; however, the inconsistent treatment protocols and different experimental designs lead to inconclusive results. Therefore, the purpose of this study is to investigate the short term and long term effect of whole body vibration on sensorimotor function in individuals with Parkinson's disease. The experimental design will be randomized double-blinded controlled trial. Sixty individuals with idiopathic Parkinson's disease will be randomly assigned to two groups and they are non-random whole body vibration group and conventional therapy group. Each participant will receive the treatment about one hour after the administration of medicine. For non-random whole body vibration group, participants will be required to maintain the erect standing position on the vibratory platform and the frequency and amplitude of vibratory stimuli will be 6Hz and 3mm respectively. Each treatment includes five sessions and each session is composed of one minute whole body vibration and one minute rest. For the conventional therapy group, participants will receive the occupational therapy including dynamic balance training and functional ambulatory training. Each session is 10 minutes in both groups and all participants will receive one and twelve treatment sessions for short-term and long-term effect respectively. Outcome measures include proprioceptive sensitivity threshold of upper limb, position sense test of the knee joint, Unified Parkinson's disease rating scale-motor (UPDRS motor), functional reach, and time up and go test (TUG). Specifically, the investigators want to answer the following four questions: 1) Is there any difference in proprioceptive sensitivity, motor performance and balance before and after treatment in individuals with Parkinson's disease? 2) Is there any difference in short-term and long term effect of whole body vibration in individuals with Parkinson's disease? 3) Is there any difference in treatment effect in individuals with Parkinson's disease in Taiwan?

ELIGIBILITY:
Inclusion Criteria:

* agree to sign the informed consent form.
* diagnosed with idiopathic Parkinson's disease with Hoehn and Yahr stage 2~3
* cognitive impairment (Mini-Mental State Examination [MMSE] score greater than 24 points
* no depression as evaluated by the Beck Depression Inventory
* no severe arm injuries or shoulder dislocation which might interfere with proprioceptive function
* can perform reaching movement
* no diagnosed peripheral nerve disorders or other neurologic conditions
* no severe tremor which might interfere with the measurement proprioceptive function

Exclusion Criteria:

* diagnosed with other central nervous system diseases, ex: stroke
* had surgeries in head or arms
* unable to sit for assessment

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change in just noticeable difference threshold of proprioceptive sensitivity | baseline, 1 day and 4 weeks
  This experiment will use psychophysical methods to assess subject perception, the psychophysical methods developed two thresholds: detection threshold/absolute threshold and difference threshold/just noticeable difference threshold (JNDT). Difference threshold represents the minimum difference between two different intensity stimulation. In this experiment, the investigator will test the difference threshold for position sense and passive motion sense
Change of position sense of the knee joint | baseline, 1 day and 4 weeks
  In the beginning, each subject sits comfortably in an arm chair (knee flexion 90o). The subject's non-affected leg is passively moved at three target angles (knee flexion 15, 30 and 70 degrees), and maintained the testing angle for 15 seconds before being return to knee flexion 90 degree (initial position). Subjects will be required to move the knee joint of the ipsilateral leg to the target angle. The assessor will use a hand-held goniometer to measure the angle of knee flexion. Each target angle will be measured three times, and both knee joints will be tested.
Change of Unified Parkinson's disease rating scale-motor (UPDRS motor) | baseline, 1 day and 4 weeks
  Unified Parkinson's disease rating scale is used to evaluate the disease progression for Parkinson's disease (PD). Higher scores represent the more advanced disease progression. It includes four subscales: mentation, behavior and mood, activities of daily living, motor examination, and complications of therapy. In this study, the investigator mainly use the motor examination subscale. There are 14 items in motor examination including speech, facial expression, tremor at test, action or postural tremor of hands, rigidity, finger taps, postural stability, gait, body bradykinesia and hypokinesia…etc. The purpose is to evaluate the motor performance for individuals with PD (Movement Disorder Society Task Force on Rating Scales for Parkinson's, 2003).
Change of balance function (measured by Functional Reach Test) | baseline, 1 day and 4 weeks
  The purpose of functional reach test is used to measure balance function. Participants can be in standing or sitting position (unable to stand). It measures the difference of distance in centimeters between arm's length with arms at 90° flexion and maximal forward reach with a fixed base of support.
Change of mobility function (measured by Time up and go test) | baseline, 1 day and 4 weeks
  The purpose of time up and go test (TUG) is to evaluate the mobility function including both static and dynamic balance. The experimenter uses a stopwatch to measure the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Participants can walk independently or with walking devices. It is easy to administer and can applied to elderly population.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou District, Taiwan

IPD SHARING:
Plan to Share IPD: No